CLINICAL TRIAL: NCT06836427
Title: CMTS0929 for Clostridioides Difficile Infection: a Prospective, Open-label, Single-arm Clinical Study
Brief Title: CMTS0929 for Clostridioides Difficile Infection
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024CMTS0929-CDI
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Clostridioides Difficile Infection
Keywords: CMTS0929; Clostridioides difficile infection; efficacy; safety
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive treatment with CMTS0929. They will be administered one unit of the liquid via colonic transendoscopic enteral tube (cTET) for three consecutive days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Eligible subjects will receive treatment with CMTS0929. They will be administered one unit of the liquid via colonic transendoscopic enteral tube (cTET) for three consecutive days.
  Interventions: Biological: CMTS0929

INTERVENTIONS:
Biological: CMTS0929 — CMTS0929 is defined as suspension from washed microbiota.

SUMMARY:
This is a prospective, open-label, single-arm study to explore the safety and the efficacy of CMTS0929 for patients with Clostridioides difficile infection (CDI).

DETAILED DESCRIPTION:
At least 12 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. Data of demographic characteristics and clinical data will be collected. After treatment, they will enter the follow-up period for safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the study:

1. At the time of informed consent, the age is between 18 and 75 years old (inclusive), including both males and non - pregnant, non - lactating females.
2. At the time of screening, meet the diagnostic criteria for Clostridioides difficile infection: a)There is a medical record proving a confirmed CDI before screening (laboratory tests show positive results for Clostridioides difficile or its toxins): positive results in Clostridioides difficile toxin detection (determined by EIAs) or colonoscopy indicating pseudomembranous colitis; or positive GDH with negative toxin results, along with obvious predisposing factors and diarrhea. b)Have an episode of CDI - related diarrhea, that is, having at least 3 bowel movements per day for at least two consecutive days and the stools are unformed (Bristol Stool Form Scale score of 6 - 7).
3. The subject or their legal representative provides informed consent, fully understands the purpose of the study, can communicate well with the researcher, and can understand and comply with all the requirements of this study.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria must be excluded from the study:

1. Subjects with immunodeficiency (such as HIV infection, or absolute neutrophil count < 0.5×10⁹/L, or total lymphocyte count < 0.5×10⁹/L, etc.), or those using immunosuppressants, or those using medium - to high - dose steroid hormones (≥20 g/d prednisone or equivalent steroid hormones).
2. Subjects with rectal outlet obstruction (such as rectal mucosal prolapse) or significant intestinal stenosis that, as evaluated by the researcher, cannot undergo cTET.
3. Before screening, subjects are diagnosed or clinically suspected of having an infection with other pathogenic microorganisms in addition to Clostridioides difficile.
4. Within 6 months before screening, subjects have undergone major abdominal surgery (excluding laparoscopic cholecystectomy or appendectomy), or have previously undergone partial or total colectomy, or partial small intestine resection, or gastroduodenal surgery.
5. At the time of screening, the subject or legal representative refuses to use effective contraceptive measures within 3 months after the last treatment.
6. As judged by the researcher, the subject is not suitable to participate in this clinical study, or participation in this clinical study cannot guarantee the rights and interests of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
The safety of CMTS0929 | Four-week
  The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0: The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.)

SECONDARY OUTCOMES:
The safety of CMTS0929 | Immediately, One-week, Two-week, Eight-week, Twenty four-week
  The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0: The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.)
The complete response rate of CDI-related diarrhea | Four-week, Eight-week
  Having no diarrhea for at least two consecutive days (with normal stool consistency (Bristol Stool Form Scale score ≤ 5) and 1-2 bowel movements per day).
The ultra-early complete response rate of CDI-related diarrhea | One-week post treatment
  Having no diarrhea for at least two consecutive days (with normal stool consistency (Bristol Stool Form Scale score ≤ 5) and 1-2 bowel movements per day).
The early complete response rate of CDI-related diarrhea | Two-week post treatment
  Having no diarrhea for at least two consecutive days (with normal stool consistency (Bristol Stool Form Scale score ≤ 5) and 1-2 bowel movements per day).
The non-response rate of CDI-related diarrhea | Two-week, Four-week, Six-week, Eight-week post treatment
  Having at least 3 bowel movements per day for at least two consecutive days and the stools are unformed (Bristol Stool Form Scale score of 6-7), and further anti-CDI treatment is required.
The recurrence rate of CDI-related diarrhea | Four-week, Six-week, Eight-week, Twenty four-week
  After the disappearance of CDI-related diarrhea, the recurrence of CDI-related diarrhea occurs, and the detection of Clostridioides difficile toxins is positive (judged by glutamate dehydrogenase [GDH] and enzyme immunoassays [EIAs]).
The major disease progression rate of CDI | Twenty four-week
  Progression to severe CDI (SCDI)/severe complicated CDI (ScCDI) (defined as high fever ≥ 38.5°C, white blood cell count > 15×10⁹/L, increased serum creatinine [> 50% higher than the baseline level], hypotension, septic shock, increased serum lactate [> 2.2 mmol/L], intestinal obstruction, toxic megacolon, intestinal perforation, or any fulminant course [i.e., the patient's condition deteriorates rapidly, or requires treatment in the intensive care unit (ICU), or is complicated by organ failure]), death, emergency colectomy, receiving ≥ 2 courses of fecal microbiota transplantation (FMT)/washed microbiota transplantation (WMT) or other forms of approved or investigational salvage therapy, or early withdrawal from the study or loss to follow-up)
The salvage/replacement treatment rate of CDI | Immediately, One-week, Two-week, Four-week, Eight-week, Twenty four-week
  The salvage/replacement treatments include receiving approved or investigational anti-infective treatment, toxin-neutralizing treatment, other FMT/WMT outside the protocol, and emergency, hospitalization, ICU or surgical treatment due to CDI-related diarrhea, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Millan B, Park H, Hotte N, Mathieu O, Burguiere P, Tompkins TA, Kao D, Madsen KL. Fecal Microbial Transplants Reduce Antibiotic-resistant Genes in Patients With Recurrent Clostridium difficile Infection. Clin Infect Dis. 2016 Jun 15;62(12):1479-1486. doi: 10.1093/cid/ciw185. Epub 2016 Mar 29. PMID 27025836
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Ng SC, Kamm MA, Yeoh YK, Chan PKS, Zuo T, Tang W, Sood A, Andoh A, Ohmiya N, Zhou Y, Ooi CJ, Mahachai V, Wu CY, Zhang F, Sugano K, Chan FKL. Scientific frontiers in faecal microbiota transplantation: joint document of Asia-Pacific Association of Gastroenterology (APAGE) and Asia-Pacific Society for Digestive Endoscopy (APSDE). Gut. 2020 Jan;69(1):83-91. doi: 10.1136/gutjnl-2019-319407. Epub 2019 Oct 14. PMID 31611298
- [Background] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878
- [Background] Ademe M. Benefits of fecal microbiota transplantation: A comprehensive review. J Infect Dev Ctries. 2020 Oct 31;14(10):1074-1080. doi: 10.3855/jidc.12780. PMID 33175698
- [Background] Drekonja D, Reich J, Gezahegn S, Greer N, Shaukat A, MacDonald R, Rutks I, Wilt TJ. Fecal Microbiota Transplantation for Clostridium difficile Infection: A Systematic Review. Ann Intern Med. 2015 May 5;162(9):630-8. doi: 10.7326/M14-2693. PMID 25938992
- [Background] Kelly CR, Fischer M, Allegretti JR, LaPlante K, Stewart DB, Limketkai BN, Stollman NH. ACG Clinical Guidelines: Prevention, Diagnosis, and Treatment of Clostridioides difficile Infections. Am J Gastroenterol. 2021 Jun 1;116(6):1124-1147. doi: 10.14309/ajg.0000000000001278. PMID 34003176
- [Background] Pike CM, Theriot CM. Mechanisms of Colonization Resistance Against Clostridioides difficile. J Infect Dis. 2021 Jun 16;223(12 Suppl 2):S194-S200. doi: 10.1093/infdis/jiaa408. PMID 33326565
- [Background] Antharam VC, Li EC, Ishmael A, Sharma A, Mai V, Rand KH, Wang GP. Intestinal dysbiosis and depletion of butyrogenic bacteria in Clostridium difficile infection and nosocomial diarrhea. J Clin Microbiol. 2013 Sep;51(9):2884-92. doi: 10.1128/JCM.00845-13. Epub 2013 Jun 26. PMID 23804381
- [Background] Guh AY, Mu Y, Winston LG, Johnston H, Olson D, Farley MM, Wilson LE, Holzbauer SM, Phipps EC, Dumyati GK, Beldavs ZG, Kainer MA, Karlsson M, Gerding DN, McDonald LC; Emerging Infections Program Clostridioides difficile Infection Working Group. Trends in U.S. Burden of Clostridioides difficile Infection and Outcomes. N Engl J Med. 2020 Apr 2;382(14):1320-1330. doi: 10.1056/NEJMoa1910215. PMID 32242357